CLINICAL TRIAL: NCT01382368
Title: Acute Effect of Sildenafil on Exercise Tolerance and Functional Capacity in COPD, IPF and Post Pneumonectomy Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Mordechai Kremer, Prof. Mordechai R. Kramer, Head of Pulmonary Institute, Rabin Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RMCBH116278 CTIL
Record Dates: First submitted 2011-05-02; First posted 2011-06-27 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; Idiopathic Pulmonary Fibrosis
Keywords: Post Pneumonectomy Patients; IPF; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Idiopathic Pulmonary Fibrosis | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sildenafil (Experimental)
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — Acute single dose of 100 mg of sildenafil. Oral intake in tablet form.

SUMMARY:
* Pulmonary diseases are increasingly important causes of morbidity and mortality in the modern world.
* Sildenafil, an orally administered a phosphodiesterase type 5 (PDE-5) inhibitor, targets the nitric oxide (NO) pathway. The drug was first approved for the treatment of Pulmonary Arterial Hypertension (PAH) in 2005.
* The aim of the suggested study is to examine the acute effect of oral intake of sildenafil on exercise tolerance and functional capacity in Chronic Obstructive Pulmonary Disease (COPD), Idiopathic pulmonary fibrosis (IPF) and post Pneumonectomy patients.
* The investigators hypothesize that oral ingestion of sildenafil prior the exercise may enhance exercise tolerance and improve function in COPD, IPF and post Pneumonectomy patients.
* Patients and Methods:

Sixty chronic lung disease patients males and females (aged 30 to 90 years) 20 COPD (GOLD III-IV) [9, 39] , 20 IPF and 20 post Pneumonectomy patients will be recruit to this study.

* All subjects will carried out two maximal cardiopulmonary exercise tests (CPET) on bicycle ergometer in different days; 60 min after intake of placebo and 60 min after intake of 100 mg sildenafil (Pfizer, Sandwich, UK), in random order.
* In first meeting prior exercise test at rest standard pulmonary function test, diffusion of CO, TLC and RV will be measured. In addition, Doppler Echocardiography and blood samples for NT-proBNP will be taken prior and post each CPET.
* After 15-20 minute of passive recovery post exercise test all patients will perform 3 short functional tests including 6 minute walk test to assess functional capacity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with severe COPD GOLD stage III- IV, FEV1 30-50% or less of predicted values, greater shortness of breath, reduced exercise capacity, repeated excretions and\ or with chronic respiratory failure [9, 39].
2. IPF patients diagnosed essentially according to the American Thoracic and European Respiratory Societies (ATS-ERS) by clinical diagnostic criteria of: (a) High-resolution computed tomography (HRCT) demonstrating a pattern of "confident" or "possible" IPF (b) Abnormal pulmonary physiology with evidence of restriction and/or impaired gas exchange (can exist during exercise alone) (c) Exclusion of other known causes of interstitial lung disease (e.g.: connective tissue disease, environmental exposure,etc.)[31].
3. Patients post Pneumonectomy more than 6 month from the amputation surgery for any diagnosis (Cancer, Trauma, and Infection- Bronchiectasis).

Exclusion Criteria:

1. Patients with known sensitivity or contraindications to phosphodiesterase 5 (PDE-5) inhibitor therapies will be excluding from the study.
2. Thromboembolic disease will be excluded by pulmonary CT-angiography or perfusion scan.
3. Patients with a history of left-sided heart failure will be excluded.
4. Patients will also exclude if they are on regular treatment with nitrates or PDE-5 inhibitors (Sildenafil, Tadalafil, Vardenafil).

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-11 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
VO2 Peak | 2-30 days between exercise tests
6 min walk test | 2-30 days between exercise tests
  Distance walked in 6 min test
Functional Tests | 2-30 days between exercise tests
  1. 30 seconds chair stand test- number of repetitions in 30 sec
  2. 8-ft-up-and -go (agility and coordination)- number of sec that takes to complete the task.

SECONDARY OUTCOMES:
Pulmonary Arterial Pressure | 2-30 days between exercise tests
NT-pro-BNP | 2-30 days between exercise tests

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai R Kramer, M.D, Principal Investigator — Rabin Medical Center, Belinson Hospital
Locations (1):
- Pulmonary Institute, Rabin Medical Center, Beilinson Hospital, Petah Tikva, Israel